CLINICAL TRIAL: NCT06974916
Title: European, Multicenter, Investigator Blinded, Randomized And Controlled Essential Tremor Trial With Staged-Bilateral FUS
Brief Title: EMBRACE Tremor BiFUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ET006
Record Dates: First submitted 2025-05-07; First posted 2025-05-16 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Essential Tremor
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Subjects will be videotaped while undergoing a standardized total CRST assessment at baseline and at the 6-month visit (use a standardized video-protocol). Subjects will wear head covers so that the investigator cannot tell whether the patient has received hair shaving to prepare for the FUS-intervention. Video-recordings will be assessed by two blinded core reviewers (i.e., certified Movement Disorder Neurologists, selected by the study Steering Committee (SC) for this task).
  The video recordings are played in random order with respect to patients and study time points to minimize reviewer bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exablate Arm (Experimental): Subjects will receive staged bilateral Exablate thalamotomy.
  Interventions: Procedure: Staged bilateral Exablate thalamotomy
- Control Arm (Active Comparator): Subjects will continue with their standard of care treatment for 6 months.
  Interventions: Other: Local standard medical treatment after previous Exablate unilateral thalamotomy.

INTERVENTIONS:
Procedure: Staged bilateral Exablate thalamotomy — Staged bilateral Exablate thalamotomy in ET patients
  Arms: Exablate Arm
Other: Local standard medical treatment after previous Exablate unilateral thalamotomy. — Local standard medical treatment
  Arms: Control Arm

SUMMARY:
This is a post-market (Phase IV) randomized, controlled, blinded, multicenter study with the aim to determine the added value of staged bilateral Exablate thalamotomy compared to a group of patients on previous unilateral treatment combined with local standard medical treatment.

DETAILED DESCRIPTION:
In patients who have undergone previous unilateral Exablate thalamotomy for Essential Tremor, the aim of this trial is to determine the effect of staged bilateral Exablate thalamotomy compared to a group of patients on previous unilateral treatment. The effect will be measured on tremor reduction, functional impairment, disease-specific quality of life, adverse events and patient-perception of the overall treatment result in patients eligible for a staged bilateral Exablate procedure.

Patients assigned to the treatment arm will receive staged bilateral Exablate thalamotomy. Patients assigned to control group will remain under local standard medical treatment.

The primary efficacy study objective is to demonstrate that Exablate staged-bilateral thalamotomy treatment reduces tremor, as measured by Treated Upper Limb CRST (A+B) (0-28) score, to a higher extent than those remaining on previous unilateral Exablate thalamotomy at 6 months.

The primary safety study objective is to assess the adverse events (AEs) of Exablate staged-bilateral thalamotomy treatment in comparison to those remaining on unilateral treatment (control group) plus medical treatment, including AE type, incidence, severity and duration at 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women with an age of 18 years or older.
2. Willing to participate in the study (i.e., signed ICF). (Willing to be randomized).
3. Patient is able to undergo a high-resolution Computerized Tomography (CT) scan.
4. Patient is able to fit into MRI unit and comply with all contraindications for the specific magnetic resonance (MR) system including and limited to contrast medium should there be needed.
5. The thalamus, sub-thalamus and the pallidum must be apparent on MR imaging.
6. Patient is able to communicate sensations to the physician during the procedure; Procedure does not require general anesthesia.
7. Patient must be able to use the Stop Sonication button freely.
8. Patient willing to have their head shaved prior to the actual treatment.
9. Patient has no history for claustrophobia which is not responding to medications.
10. ET patients who are eligible for second side staged bilateral Exablate thalamotomy treatment. Time since first intervention is at least 9 months.
11. Available tremor assessment prior to the unilateral Exablate thalamotomy.
12. Patients randomized to the study, irrespective of group allocation should be willing and able to remain in the study for at least 6 months and able to complete the required assessments.

Exclusion Criteria:

1. Subject experienced any non-transient neurological event or worsening following the previous Exablate procedure.
2. Patients with MRI related contraindications (e.g. presence of metallic implants incompatibility with MRI, severe claustrophobia, reaction to contrast medium).
3. Patients in whom it is not possible to avoid energy absorbing structures or sensitive tissues (e.g., skull implants, surgical clips, shunts, electrodes, dura patch, skull patch, electrodes, etc.) from the path of the ultrasound beam.
4. Patients with concurrent active infections disease and/or severe allergies with fever.
5. Patients that have been diagnosed with brain tumors or a vascular anomaly.
6. Patients with a history of seizures, brain hemorrhages, stroke within the past year, or any coagulopathy.
7. Patients under anticoagulants and/or anti-platelets drugs known to increase bleeding risk within the duration defined by the half-life of the specific drugs.
8. Patient that has been given any contrast agent (e.g., CT, MRI), within 24 hours before treatment
9. Severe unstable hypertension that cannot be controlled by medications (diastolic Blood Pressure > 100 on medication).
10. Patients with unstable cardiac status.
11. Patients exhibiting any behavior(s) consistent with ethanol or substance abuse.
12. Cerebrovascular disease (multiple CVA or CVA within 6 months).
13. Patients with risk factors for intraoperative or postoperative bleeding.
14. Imaging shows abnormal finding in CT or/and MRI (e.g., brain tumor, brain vascular malformation, shunt, etc.).
15. Patient has physical subscale score ≥ 16.5 on the Dysphagia Handicap Index or has been diagnosed with dysphagia.
16. Patient with cognitive impairment.
17. Patient with clinically significant abnormal speech function as determined by a speech pathologist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Treated Upper Limb Clinical Rating Scale for Tremor (CRST) (A+B) (0-28) score for the treated side. | 6 Months
  The primary endpoint is the difference of the Treated Upper Limb CRST (A+B) score between groups at 6 months. Higher score means a worse tremor.

SECONDARY OUTCOMES:
Treated Upper Limb Clinical Rating Scale for Tremor (CRST) (A+B) (0-28) score as assessed by the blinded reviewers of the video-recordings. | 6 Months, 12 Months
  Between group comparison through month 6 and within group comparison vs baseline up to month 12 in Treated Upper Limb CRST (A+B) score as assessed by the blinded reviewers of the video-recordings. Higher score means a worse tremor.
Clinical Rating Scale for Tremor (CRST) part A (0-76) | 6 Months, 12 Months
  Between group comparison through month 6 and within group comparison vs baseline up to month 12 in resting, postural, and action tremors of all items as measured by CRST part A. Higher score means a worse tremor.
Bilateral Upper Limb Clinical Rating Scale for Tremor (CRST) (A+B) (0-56) | 6 Months, 12 Months
  Between group comparison through month 6 and within group comparison vs baseline up to month 12 in Bilateral Upper Limb CRST (A+B). Higher score means a worse tremor.
Total Clinical Rating Scale for Tremor (CRST) (A+B) (0-116) | 6 Months, 12 Months
  Between group comparison through month 6 and within group comparison vs baseline up to month 12 in Total CRST (A+B). Higher score means a worse tremor.
Clinical Rating Scale for Tremor (CRST) part C (0-32) | 6 Months, 12 Months
  Between group comparison through month 6 and within group comparison vs baseline up to month 12 in functional disabilities as measured by CRST part C. Higher score means a worse tremor.
Axial Clinical Rating Scale for Tremor (CRST) (0-20) | 6 Months, 12 Months
  Between group comparison through month 6 and within group comparison vs baseline up to month 12 in Axial CRST defined as face, tongue, head tremor and voice items of CRST part A
Quality of life questionnaire | 6 Months, 12 Months
  Between group comparison through month 6 and within group comparison vs baseline up to month 12 in disease specific QOL
Change of tremor medication | 6 Months, 12 Months
  Between group comparison through month 6 and within group comparison vs baseline up to month 12 in tremor medication change
Safety: Incidence and frequency of adverse events related to the treatment. | 6 Months, 12 Months
  Incidence and frequency of adverse events related to the treatment and/or procedure. The investigator will capture any untoward events in the case report forms along with severity, duration, and resolution, and whether the event is considered serious. The severity of adverse events will be categorized according to the definition of adverse events from the International Organization for Standardization (ISO).

OTHER OUTCOMES:
Objective assessment of specific adverse events | 6 Months, 12 Months
  Objective assessment of specific adverse events will be carried out for Speech, Gait and Motor Strength at baseline and 6 months and eventually at 12 months. If the adverse reported in the objective assessment is resolved at 6 months (Speech, Gait and Motor strength) it will not be carried out for the 12-month visit.
Patient Global Impression of Change (PGIC) | 6 Months, 12 Months
  Between group comparison through month 6 and within group comparison vs baseline up to month 12 in Patient Global Impression of Change (PGIC). PGIC is a 7-point scale depicting a patient's rating of overall improvement. Higher score means a worse condition.
Clinician Global Impression of Change (CGIC) | 6 Months, 12 Months
  Between group comparison through month 6 and within group comparison vs baseline up to month 12 in Clinician Global Impression of Change (CGIC). The CGIC comprises two companion one-item measures evaluating the following: (a) severity of pathology from 1 to 7 and (b) change from the initiation of treatment on a similar seven-point scale. Higher score means a worse condition.
Caregiver Global Impression of Change (CaGIC) | 6 Months, 12 Months
  Between group comparison through month 6 and within group comparison vs baseline up to month 12 in Caregiver Global Impression of Change (CaGIC). The CaGIC comprises two companion one-item measures evaluating the following: (a) severity of pathology from 1 to 7 and (b) change from the initiation of treatment on a similar seven-point scale. Higher score means a worse condition.
Responder analysis | 6 Months
  A responder analysis will be performed to compute the proportion of subjects achieving a clinically satisfactory result. The CRST will be used. The responder analysis will be based on this scoring:
  * Full responder: no tremor (0) or barely no tremor (1).
  * Partial responder: moderate tremor, < 2cm, (2)
  * Insufficient responder: marked (2-4 cm, 3) or severe (> 4 cm)

CONTACTS AND LOCATIONS:
Overall Officials: Günther Deuschl, Principal Investigator — Universitätsklinikum Schleswig-Holstein, Campus Kiel (UKSH); Steffen Paschen, Principal Investigator — Universitätsklinikum Schleswig-Holstein, Campus Kiel (UKSH)
Locations (6):
- Turku University Hospital, Turku, Finland
- Universitätsklinikum Schleswig-Holstein, Campus Kiel (UKSH), Kiel, Germany
- Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan, Italy
- Spain (3):
  - Germans Trias i Pujol Hospital, Badalona
  - HM CINAC- Hospital Universitario HM Puerta del Sur, Móstoles
  - Clinica Universidad de Navarra, Pamplona

IPD SHARING:
Plan to Share IPD: No